CLINICAL TRIAL: NCT06400589
Title: A Phase 3, Multicenter, Randomized, Double-Masked and Vehicle-Controlled Study Evaluating the Efficacy and Safety of Tanfanercept (HL036) Ophthalmic Solution 0.25% and 1.0% Compared to Vehicle in Participants With Dry Eye Disease (VELOS-4)
Brief Title: A Study to Evaluate the Efficacy and Safety of Tanfanercept (HL036) in Dry Eye Disease
Acronym: VELOS-4
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Logistical issue
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HL036-DED-US-P303
Record Dates: First submitted 2024-04-29; First posted 2024-05-06 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.25% tanfanercept (Experimental): 0.25% tanfanercept ou bid for 12 weeks
  Interventions: Drug: tanfanercept
- 1.0% tanfanercept (Experimental): 1.0% tanfanercept ou bid for 12 weeks
  Interventions: Drug: tanfanercept
- Vehicle (Placebo Comparator): Vehicle ou bid for 12 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: tanfanercept — TNF inhibitor
  Arms: 0.25% tanfanercept; 1.0% tanfanercept
Drug: Vehicle — Same composition as tanfanercept but without the active ingredient
  Arms: Vehicle

SUMMARY:
The objectives of this study are to compare the efficacy and safety of tanfanercept ophthalmic solution 0.25% and 1.0% to vehicle for the treatment of DED.

DETAILED DESCRIPTION:
The purpose of this research study is to test the safety and effectiveness (how well the drug works) of Tanfanercept ophthalmic solution 0.25% and Tanfanercept ophthalmic solution 1% against vehicle (no active treatment). Effectiveness will be measured by the improvement in Schirmer Test results (a test to see how many tears you produce), reduction of dry eye symptoms, eye redness (conjunctival redness), and eye surface irritation (corneal staining, conjunctival staining). Eye safety assessments will also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years of age
2. Provide written informed consent
3. Are willing to attend all study visits and able to comply with study procedures and assessments
4. Have a self-reported history of DED (OU) for at least 6 months prior to Visit 1

Exclusion Criteria:

1. Have an uncontrolled systemic disease
2. Have been exposed to an investigational drug or device within 30 days or 5 half-lives prior to Visit 1, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Schirmer Test | 12 weeks
  The proportion of participants with improvement from baseline in unanesthetized Schirmer

SECONDARY OUTCOMES:
Schirmer Test | 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Change from baseline in unanesthetized Schirmer test score
Symptom Assessment in Dry Eye | 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Change from baseline in Symptom Assessment in Dry Eye
VAS | 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Change from baseline in Eye dryness, burning/stinging, itching, foreign body sensation, eye discomfort, photophobia, and pain on the visual analog scale (VAS)
Conjunctival redness | 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Change from baseline in conjunctival redness on BHVI bulbar redness scale
Corneal staining | 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Change from baseline in corneal staining on NEI scale

OTHER OUTCOMES:
Comfort Score (Exploratory) | 2 weeks, 4 weeks, 8 weeks
  Study product instillation score at each post-baseline visit

CONTACTS AND LOCATIONS:
Locations (1):
- HanAll Site #1, Delray Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No